CLINICAL TRIAL: NCT02680665
Title: AMEPAROMO CAPSULES 250 MG DRUG USE INVESTIGATION
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3391001
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Intestinal Amebiasis
MeSH Terms: conditions — Dysentery, Amebic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This Study is intended to evaluate the safety and effectiveness of Ameparomo Capsules 250 mg under actual medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no history of using this product

Exclusion Criteria:

* No exclusion criteria are set out in this study.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sites of infection department, internal medicine, and other relevant departments.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3391001&StudyName=Drug%20Use%20Investigation%20Of%20Paromomycin.%20%28regulatory%20Post%20Marketing%20Commitment%20Plan%29.

RESULTS

PARTICIPANT FLOW:
Groups:
- AMEPAROMO Capsules (Paromomycin): Participants who received AMEPAROMO capsules as indicated in the approved local product document were observed for a period of 10 days at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | AMEPAROMO Capsules (Paromomycin)
Started | 120
Completed | 115
Not Completed | 5
Not completed — No visit after the first prescription | 5

BASELINE CHARACTERISTICS:
Population: A total of 120 participants were enrolled in this study. Of the 120 participants, 5 participants were excluded from the safety analysis set due to following reasons: no visit after the first prescription day (n=5).
Arm/Group | AMEPAROMO Capsules (Paromomycin)
Number analyzed (Participants) | 115
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 to <65 years | 100
  ≥ 65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to AMEPAROMO capsules in a participant who received AMEPAROMO capsules. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to AMEPAROMO capsules was assessed by the physician.
Time Frame: 38 days at maximum
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received AMEPAROMO capsules at least once.
Measure: Number; unit: Particpants
Arm/Group | AMEPAROMO Capsules (Paromomycin)
Number analyzed (Participants) | 115
Particpants
  ADRs | 15
  Serious ADRs | 0

2. Secondary Outcome: Proportion of Cyst Negative
Description: Proportion of cyst negative, which was defined as the percentage of participants with negative results in the examination of cysts after AMEPAROMO capsules up to 3 months after the completion of observation period or discontinuation of treatment, was presented along with its 2-sided 95% CI. The results of the examination of cysts were assessed as "negative ", "positive", or "indeterminate".
Time Frame: 10 days + 3 months at maximum
Population: The cyst analysis set consists of the participants in the safety analysis set who have undergone the cyst examination at the end of the observation period or at the time of treatment discontinuation. Participants with no information on cyst examination (53) and those with non-target disease (9) were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | AMEPAROMO Capsules (Paromomycin)
Number analyzed (Participants) | 53
Percentage of Participants | 98.1 [89.9 to 100.0]

3. Secondary Outcome: Overall Clinical Response Rate
Description: Clinical response rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with its 2-sided 95% CI. Clinical response of AMEPAROMO capsules was assessed as "effective", "not effective", or "indeterminate" by the physician based on the clinical course at the end of the observation period or at the time of treatment discontinuation.
Time Frame: 10 days at maximum
Population: The clinical response analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at the end of the observation period or at the time of treatment discontinuation. Participants with non-target disease (9) and participants who assessed as indeterminate at the final observation (6) were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | AMEPAROMO Capsules (Paromomycin)
Number analyzed (Participants) | 100
Percentage of Participants | 99.0 [94.6 to 100.0]

ADVERSE EVENTS:
Time Frame: 38 days at maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | AMEPAROMO Capsules (Paromomycin)
All-Cause Mortality (participants affected / at risk) | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115
Other Adverse Events (participants affected / at risk) | 18/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMEPAROMO Capsules (Paromomycin) (N=115)
Diarrhoea (Gastrointestinal disorders) | 15 — Diarrhoea
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT02680665/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02680665/SAP_001.pdf